CLINICAL TRIAL: NCT04346706
Title: Radiographic Evaluation of Marginal Bone Level, Buccal and Palatal Plate Thickness Alteration, and Implant Stability After Placement in Healed Ridges and Fresh Extraction Sockets: A 6 Months Prospective Study.
Brief Title: Immediate Implant Placement in Fresh Extraction Sockets and Delayed Implants in Healed Sockets.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Nada BOU ABBOUD NAAMAN, Principal investigator, Saint-Joseph University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMD124
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Tooth Extraction; Dental Implantation; Bone Remodeling
Keywords: Dental implantation; Immediate dental implant loading; Marginal bone remodeling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiographic measurements were done by a different clinician than the surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implantation (Experimental): Tooth extraction, immediate insertion of an implant with immediate temporization
  Interventions: Device: Extraction and Implant insertion (test)
- Delayed implantation (Experimental): Implant inserted in a healed socket with immediate temporization
  Interventions: Device: Implant insertion (control)

INTERVENTIONS:
Device: Extraction and Implant insertion (test) — The surgical procedure was conducted under local anesthesia. Intrasulcular incisions were performed around the mesial and distal tooth to the implant recipient site. Buccal and palatal mucoperiosteal flaps were elevated. Tooth extractions were carried out atraumatically using periotomes. Implant site preparation was completed in compliance with the general surgical principles and protocols defined by the manufacturer and screw-shaped implants (UFII, DIO™) were inserted at no less than 35 Ncm. Final insertion torque (IT) was measured and recorded using a manual hand wrench (DIO™). Resonance frequency analysis (RFA) was performed using an Osstell device (Sävedalen, Sweden). For each implant, three Implant Stability Quotient (ISQ) readings were recorded by the same operator to calculate the mean ISQ, at implant placement (T0) and 3 months after implant insertion (T3) prior to final abutment torque and crown cementation.
  Absorbable interrupted 4.0 sutures were used for flap closure.
  Arms: Immediate implantation
Device: Implant insertion (control) — The surgical procedure was conducted under local anesthesia. Intrasulcular incisions were performed around the mesial and distal tooth to the implant recipient site. Buccal and palatal mucoperiosteal flaps were elevated, the implant site preparation was completed in compliance with the general surgical principles and protocols defined by the manufacturer and screw-shaped implants (UFII, DIO™) were inserted at no less than 35 Ncm. Final insertion torque (IT) was measured and recorded using a manual hand wrench (DIO™). Resonance frequency analysis (RFA) was performed using an Osstell device (Sävedalen, Sweden). For each implant, three Implant Stability Quotient (ISQ) readings were recorded by the same operator to calculate the mean ISQ. This was done at implant placement (T0) and 3 months after implant insertion (T3) prior to final abutment torque and crown cementation.
  Absorbable interrupted 4.0 sutures were used for flap closure.
  Arms: Delayed implantation

SUMMARY:
The purpose of this prospective clinical study was to compare in delayed and immediately placed implants, the marginal vertical bone loss at 4 sides of the implant (buccal, palatal, mesial and distal), as well as the buccal and palatal bone thickness reduction at 3 months after loading.

DETAILED DESCRIPTION:
Twenty-four patients were consecutively selected and enrolled in this study based on the aforementioned exclusion and inclusion criteria. Clinical examination was done by a different clinician than the operator, and according to the treatment indication, patients were allocated to the delayed implant placement group (Control), or the immediate implant placement group (Test). Thus, 15 implants were placed in healed extraction sites and immediately temporized (Control group), and 15 implants were placed in immediate extraction sites with immediate temporization (Test group).

Provisional acrylic crowns were prepared. All patients were placed on a prophylactic antibiotic regimen, starting one day prior to surgery as they were asked to take amoxicillin 500 mg; three times a day for 10 days or clindamycin 300 mg twice daily for 10 days for penicillin-allergic patients.

For the test group, tooth extractions were carried out atraumatically using periotomes. In both groups, the implant site preparation was completed in compliance with the general surgical principles and protocols defined by the manufacturer and screw-shaped implants (UFII, DIO™) were inserted at no less than 35 Ncm.

Temporary abutments were connected to the implants and torqued at 20 Ncm, and then temporary crowns were cemented on top of the abutments after checking and reducing occlusion to non-existent in both centric and lateral excursions.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old, compliant (willing to show up to all their follow-up visits), and able to read, understand and sign an informed consent. All patients were to have good oral hygiene levels (full mouth plaque scores (FMPS) <15-20%, and full mouth bleeding index (FMBI) <15-20%), requiring implant insertion in a maxillary premolar site either immediately or in a healed "pristine bone".

Exclusion Criteria:

* Presence of major contraindications to implant surgery, patients that had received head and neck radiation for cancer treatment, immunosuppressed or immunocompromised patients, uncontrolled diabetes, pregnant or breast-feeding woman, untreated periodontitis and/or poor oral hygiene and motivation, presence of buccal dehiscence, and finally previous bone grafting or ridge preservation in the studied area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline of marginal vertical bone level at 6 months | Following procedure at day 0 (implant insertion) and 6 months (post-implantation)
  Marginal vertical bone level changes at 4 sides of the implant (buccal, palatal, mesial and distal) on Cone Beam Computed Tomography (CBCT) images
Change from baseline of bone plate thickness at 6 months | Following procedure at day 0 (implant insertion) and 6 months (post-implantation)
  Buccal and palatal bone thickness at 4 levels : 0 mm, 2 mm, 4 mm and 6 mm from the implant platform on CBCT images

SECONDARY OUTCOMES:
Change from baseline of implant stability quotient at 3 months | Following procedure at day 0 (implant insertion) and 3 months (post-implantation)
  Measurements of implant stability quotient (ISQ) following implant insertion
Record of insertion torque | Following procedure at day 0 (implant insertion)
  Insertion torque value at implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Nada Naaman, PhD, Study Director — Saint-Joseph University
Locations (1):
- Saint-Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Patient characteristics. Outcome measures
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication for 10 years
Access Criteria: The complete dataset can be available for researchers working on a meta-analysis

REFERENCES:
- [Background] Penarrocha-Diago M, Demarchi CL, Maestre-Ferrin L, Carrillo C, Penarrocha-Oltra D, Penarrocha-Diago MA. A retrospective comparison of 1,022 implants: immediate versus nonimmediate. Int J Oral Maxillofac Implants. 2012 Mar-Apr;27(2):421-7. PMID 22442783
- [Background] Kim JK, Yoon HJ. Clinical and radiographic outcomes of immediate and delayed placement of dental implants in molar and premolar regions. Clin Implant Dent Relat Res. 2017 Aug;19(4):703-709. doi: 10.1111/cid.12496. Epub 2017 May 18. PMID 28517552
- [Background] Atieh MA, Alsabeeha NH, Duncan WJ, de Silva RK, Cullinan MP, Schwass D, Payne AG. Immediate single implant restorations in mandibular molar extraction sockets: a controlled clinical trial. Clin Oral Implants Res. 2013 May;24(5):484-96. doi: 10.1111/j.1600-0501.2011.02415.x. Epub 2012 Jan 26. PMID 22276690
- [Background] Mello CC, Lemos CAA, Verri FR, Dos Santos DM, Goiato MC, Pellizzer EP. Immediate implant placement into fresh extraction sockets versus delayed implants into healed sockets: A systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2017 Sep;46(9):1162-1177. doi: 10.1016/j.ijom.2017.03.016. Epub 2017 May 3. PMID 28478869
- [Background] Lindeboom JA, Tjiook Y, Kroon FH. Immediate placement of implants in periapical infected sites: a prospective randomized study in 50 patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Jun;101(6):705-10. doi: 10.1016/j.tripleo.2005.08.022. Epub 2006 Mar 22. PMID 16731387
- [Background] Rowan M, Lee D, Pi-Anfruns J, Shiffler P, Aghaloo T, Moy PK. Mechanical versus biological stability of immediate and delayed implant placement using resonance frequency analysis. J Oral Maxillofac Surg. 2015 Feb;73(2):253-7. doi: 10.1016/j.joms.2014.09.024. Epub 2014 Oct 13. PMID 25579008
- [Background] Esposito M, Zucchelli G, Cannizzaro G, Checchi L, Barausse C, Trullenque-Eriksson A, Felice P. Immediate, immediate-delayed (6 weeks) and delayed (4 months) post-extractive single implants: 1-year post-loading data from a randomised controlled trial. Eur J Oral Implantol. 2017;10(1):11-26. PMID 28327692
- [Background] Berberi AN, Sabbagh JM, Aboushelib MN, Noujeim ZF, Salameh ZA. A 5-year comparison of marginal bone level following immediate loading of single-tooth implants placed in healed alveolar ridges and extraction sockets in the maxilla. Front Physiol. 2014 Jan 31;5:29. doi: 10.3389/fphys.2014.00029. eCollection 2014. PMID 24550840
- [Background] Buser D, Janner SF, Wittneben JG, Bragger U, Ramseier CA, Salvi GE. 10-year survival and success rates of 511 titanium implants with a sandblasted and acid-etched surface: a retrospective study in 303 partially edentulous patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):839-51. doi: 10.1111/j.1708-8208.2012.00456.x. PMID 22897683
- [Background] Ostman PO, Hellman M, Sennerby L. Ten years later. Results from a prospective single-centre clinical study on 121 oxidized (TiUnite) Branemark implants in 46 patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):852-60. doi: 10.1111/j.1708-8208.2012.00453.x. Epub 2012 May 29. PMID 22642261
- [Background] Romeo E, Lops D, Margutti E, Ghisolfi M, Chiapasco M, Vogel G. Long-term survival and success of oral implants in the treatment of full and partial arches: a 7-year prospective study with the ITI dental implant system. Int J Oral Maxillofac Implants. 2004 Mar-Apr;19(2):247-59. PMID 15101597
- [Background] Covani U, Chiappe G, Bosco M, Orlando B, Quaranta A, Barone A. A 10-year evaluation of implants placed in fresh extraction sockets: a prospective cohort study. J Periodontol. 2012 Oct;83(10):1226-34. doi: 10.1902/jop.2012.110583. Epub 2012 Jan 5. PMID 22220768
- [Background] Fugazzotto PA. Implant placement at the time of mandibular molar extraction: description of technique and preliminary results of 341 cases. J Periodontol. 2008 Apr;79(4):737-47. doi: 10.1902/jop.2008.070293. PMID 18380569
- [Background] Gher ME, Quintero G, Assad D, Monaco E, Richardson AC. Bone grafting and guided bone regeneration for immediate dental implants in humans. J Periodontol. 1994 Sep;65(9):881-91. doi: 10.1902/jop.1994.65.9.881. PMID 7990026
- [Background] Schwartz-Arad D, Chaushu G. Placement of implants into fresh extraction sites: 4 to 7 years retrospective evaluation of 95 immediate implants. J Periodontol. 1997 Nov;68(11):1110-6. doi: 10.1902/jop.1997.68.11.1110. PMID 9407405
- [Background] Atsumi M, Park SH, Wang HL. Methods used to assess implant stability: current status. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):743-54. PMID 17974108
- [Background] Meredith N, Shagaldi F, Alleyne D, Sennerby L, Cawley P. The application of resonance frequency measurements to study the stability of titanium implants during healing in the rabbit tibia. Clin Oral Implants Res. 1997 Jun;8(3):234-43. doi: 10.1034/j.1600-0501.1997.080310.x. PMID 9586468
- [Background] Orlando B, Barone A, Giorno TM, Giacomelli L, Tonelli P, Covani U. Insertion torque in different bone models with different screw pitch: an in vitro study. Int J Oral Maxillofac Implants. 2010 Sep-Oct;25(5):883-7. PMID 20862400
- [Background] Zimmermann J, Sommer M, Grize L, Stubinger S. Marginal bone loss 1 year after implantation: a systematic review for fixed and removable restorations. Clin Cosmet Investig Dent. 2019 Jul 16;11:195-218. doi: 10.2147/CCIDE.S208076. eCollection 2019. PMID 31406478
- [Background] Galindo-Moreno P, Leon-Cano A, Ortega-Oller I, Monje A, O Valle F, Catena A. Marginal bone loss as success criterion in implant dentistry: beyond 2 mm. Clin Oral Implants Res. 2015 Apr;26(4):e28-e34. doi: 10.1111/clr.12324. Epub 2014 Jan 3. PMID 24383987
- [Background] Vignoletti F, Sanz-Esporrin J, Sanz-Martin I, Nunez J, Luengo F, Sanz M. Ridge alterations after implant placement in fresh extraction sockets or in healed crests: An experimental in vivo investigation. Clin Oral Implants Res. 2019 Apr;30(4):353-363. doi: 10.1111/clr.13421. Epub 2019 Apr 3. PMID 30864234
- [Background] Juodzbalys G, Wang HL. Esthetic index for anterior maxillary implant-supported restorations. J Periodontol. 2010 Jan;81(1):34-42. doi: 10.1902/jop.2009.090385. PMID 20059415
- [Background] Buser D, Wittneben J, Bornstein MM, Grutter L, Chappuis V, Belser UC. Stability of contour augmentation and esthetic outcomes of implant-supported single crowns in the esthetic zone: 3-year results of a prospective study with early implant placement postextraction. J Periodontol. 2011 Mar;82(3):342-9. doi: 10.1902/jop.2010.100408. Epub 2010 Sep 10. PMID 20831371
- [Background] Esposito M, Klinge B, Meyle J, Mombelli A, Rompen E, van Steenberghe D, Van Dyke T, Wang HL, van Winkelhoff AJ. Working Group on the Treatment Options for the Maintenance of Marginal Bone Around Endosseous Oral Implants, Stockholm, Sweden, 8 and 9 September 2011. Consensus statements. Eur J Oral Implantol. 2012;5 Suppl:S105-6. No abstract available. PMID 22834399
- [Background] Ormianer Z, Piek D, Livne S, Lavi D, Zafrir G, Palti A, Harel N. Retrospective clinical evaluation of tapered implants: 10-year follow-up of delayed and immediate placement of maxillary implants. Implant Dent. 2012 Aug;21(4):350-6. doi: 10.1097/ID.0b013e31825feb16. PMID 22814562
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Background] Tarnow DP, Cho SC, Wallace SS. The effect of inter-implant distance on the height of inter-implant bone crest. J Periodontol. 2000 Apr;71(4):546-9. doi: 10.1902/jop.2000.71.4.546. PMID 10807116
- [Background] Hermann JS, Cochran DL, Nummikoski PV, Buser D. Crestal bone changes around titanium implants. A radiographic evaluation of unloaded nonsubmerged and submerged implants in the canine mandible. J Periodontol. 1997 Nov;68(11):1117-30. doi: 10.1902/jop.1997.68.11.1117. PMID 9407406
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Puisys A, Auzbikaviciute V, Minkauskaite A, Simkunaite-Rizgeliene R, Razukevicius D, Linkevicius R, Linkevicius T. Early crestal bone loss: Is it really loss? Clin Case Rep. 2019 Aug 27;7(10):1913-1915. doi: 10.1002/ccr3.2376. eCollection 2019 Oct. PMID 31624607
- [Background] O'Sullivan D, Sennerby L, Jagger D, Meredith N. A comparison of two methods of enhancing implant primary stability. Clin Implant Dent Relat Res. 2004;6(1):48-57. doi: 10.1111/j.1708-8208.2004.tb00027.x. PMID 15595709
- [Background] Nedir R, Bischof M, Szmukler-Moncler S, Bernard JP, Samson J. Predicting osseointegration by means of implant primary stability. Clin Oral Implants Res. 2004 Oct;15(5):520-8. doi: 10.1111/j.1600-0501.2004.01059.x. PMID 15355393
- [Background] Lages FS, Douglas-de Oliveira DW, Costa FO. Relationship between implant stability measurements obtained by insertion torque and resonance frequency analysis: A systematic review. Clin Implant Dent Relat Res. 2018 Feb;20(1):26-33. doi: 10.1111/cid.12565. Epub 2017 Dec 1. PMID 29194944
- [Background] Berglundh T, Lindhe J. Healing around implants placed in bone defects treated with Bio-Oss. An experimental study in the dog. Clin Oral Implants Res. 1997 Apr;8(2):117-24. doi: 10.1034/j.1600-0501.1997.080206.x. PMID 9758962
- [Background] Lee DW, Choi YS, Park KH, Kim CS, Moon IS. Effect of microthread on the maintenance of marginal bone level: a 3-year prospective study. Clin Oral Implants Res. 2007 Aug;18(4):465-70. doi: 10.1111/j.1600-0501.2007.01302.x. Epub 2007 Apr 18. PMID 17441983
- [Derived] Dagher M, Mokbel N, Aboukhalil R, Ghosn N, Kassir A, Naaman N. Marginal Bone Level and Bone Thickness Reduction in Delayed and Immediate Implant Placement Protocol 6 Months Post-loading: An Observational Clinical Prospective Study. J Maxillofac Oral Surg. 2022 Jun;21(2):571-579. doi: 10.1007/s12663-021-01673-3. Epub 2022 Jan 7. PMID 35712433